CLINICAL TRIAL: NCT03769805
Title: Clinical Study of Anlotinib in Maintenance Treatment of Advanced NSCLC
Acronym: CSOAIMTOAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Huai'an First People's Hospital (Other); Jiangsu Taizhou People's Hospital (Other); Zhongda Hospital (Other); Yancheng City NO.1 People's Hospital (Unknown); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L014
Record Dates: First submitted 2018-11-26; First posted 2018-12-10 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Nonsmall Cell Lung Cancer
Keywords: anlotinib; Maintenance treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Arm (Experimental): Anlotinib hydrochloride capsule 12 mg, orally, once a day, oral before breakfast, according to the research program for 2 weeks, discontinued for 1 week. Patients with complete remission (CR), partial remission (PR) and stable disease (SD) continued to administer drugs until the disease progressed, intolerable toxicity or withdrawal was required. Patients with progression of illness (PD) discontinued their medication.
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib hydrochloride capsule 12 mg, orally, once a day, oral before breakfast, according to the research program for 2 weeks, discontinued for 1 week.

SUMMARY:
Based on the need of clinical practice of maintenance therapy for advanced NSCLC and the reliable data of third-line treatment for non-small cell lung cancer, the investigators designed a clinical study of antinil hydrochloride versus pemetrexed in maintenance therapy for advanced NSCLC to prospectively evaluate the efficacy of antinil hydrochloride in maintenance therapy for advanced NSCLC. Value, to provide a scientific basis for prolonging the survival time of patients with advanced NSCLC, improving the quality of life of patients in the course of treatment, and optimizing treatment strategies to a greater extent.

DETAILED DESCRIPTION:
This study is planned to be carried out in Jiangsu regional multi-center. 83 cases are preliminarily expected to be included. The study started in December 2018 and ended in December 2019. It is expected that the trial will end in December 2020.

In the absence of such situations as withdrawal of informed consent, intolerance of drug toxicity and side effects, or inappropriateness for further trials, each participant's expected time for research and treatment will continue until radiographically confirmed tumor progression occurs.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC was diagnosed by cytology or histology, and patients with stage IIIB or IV and no sensitive mutation of EGFR/ALK/ROS1 were diagnosed according to IASLC Staging Standard (IASLC 2007 9) of the 7th edition of 2009;
* Those who had received platinum-containing two-drug combination chemotherapy for 4-6 cycles were judged as complete remission (CR), partial remission (PR) and stabilization (SD) according to RECIST 1.1 standard; (Specific schemes of platinum-containing two-drug combination chemotherapy included vinorelbine+cisplatin/carboplatin, gemcitabine+cisplatin/carboplatin, paclitaxel+cisplatin/carboplatin, albumin. Binding paclitaxel + cisplatin / carboplatin, docetaxel + cisplatin / carboplatin, pemetrexed + cisplatin / carboplatin, and squamous cell carcinoma may include docetaxel + nedaplatin)
* Age: 18 to 74 years old, regardless of gender;
* PS 0～1(ECOG) ;
* The life expectancy is more than 3 months;
* According to RECIST 1.1 criteria, patients have at least one imaging (CT, MRI) lesion that can be measured or evaluated; the lesion was not previously treated by radiotherapy. The longest diameter of the target lesion should be greater than or equal to 10 mm (the short axis of lymph node is greater than or equal to 15 mm);
* Patients with brain metastasis at baseline should be single intracranial metastasis, asymptomatic or asymptomatic after treatment;
* Women: For all women who may be pregnant, pregnancy tests must be performed within 72 hours before starting treatment, or medically approved contraceptive methods must be used within three months after the treatment and during the period after the end of treatment; serum or urine pregnancy tests must be negative and must be non-lactating; Male: Contraceptive measures were taken during and within 3 months after surgical sterilization or treatment;
* The functional level of organs must meet the following requirements:

Routine blood test ANC is more than 1.5 x 109/L; PLT is more than 90 x 109/L; Hb > 90g/L Blood biochemistry TBIL is less than 1.5 x ULN ALT and AST < 2 *ULN; for patients with liver metastases, ALT and AST < 5 *ULN; BUN and CR were less than 1.5 x ULN and creatinine clearance was more than 50 ml/min.

Colour Sonography LVEF is more than 50%; 12 lead electrocardiogram The Fridericia-corrected QTcF was < 450 ms for males and < 470 MS for females.

* Subjects who have the ability to understand and sign the informed consent must sign the informed consent before any screening evaluation.

Exclusion Criteria:

* Unable to swallow, chronic diarrhea and intestinal obstruction, there are many factors affecting drug use and absorption;
* There is a third interstitial effusion (e.g. massive pleural and ascites) that cannot be controlled by drainage or other means;
* Radiotherapy, surgical treatment, or other targeted therapy for non-small cell lung cancer was given within four weeks before the first study drug was administered;
* Researchers judged that they had not recovered from previous adverse events before taking the drug for the first time (NCI-CTCAE Version 4.0 Grade > Grade 1);
* Patients with multiple or active (uncontrolled) brain metastases, cancerous meningitis, spinal cord compression, or with brain or pia mater diseases detected by CT or MRI at screening time (patients with single brain metastases whose symptoms were stable and had completed treatment within 28 days prior to the first use of the research drug) may be enrolled in the group, but only through craniocerebral MRI, CT or venography. Shadow evaluation confirmed no symptoms of cerebral hemorrhage;
* Participated in other drug clinical trials within 4 weeks before taking the first research drug;
* There was a history of bleeding. Within 4 weeks before screening, any bleeding events with a severe grade of 3 or more in CTCAE 4.0 occurred;
* Having a history of thrombosis, or judging by researchers, abnormal coagulation function has clinical significance, tends to bleed, or is undergoing thrombolysis or anticoagulation therapy;
* Hemoptysis was evident within 2 months before the first study drug was administered;
* Patients with hypertension who could not be well controlled by a single antihypertensive drug (systolic pressure > 140 mmHg, diastolic pressure > 90 mmHg); patients with a history of unstable angina pectoris; newly diagnosed angina pectoris in the first three months of screening or myocardial infarction events in the first six months of screening; arrhythmia (including QTcF: males > 450 ms, females) Long-term use of antiarrhythmic drugs and New York Heart Association Classification (> Class II) cardiac insufficiency were required;
* Urinary routine indicated that urinary protein (++) and confirmed 24-hour urinary protein quantification > 1.0 G;
* Long-term union of wounds or incomplete healing of fractures;
* Other malignant tumors in the past five years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma;
* Those with allergic constitution or known history of allergy to the drug components of this regimen;
* Has a history of immunodeficiency, including HIV positive testing, or other acquired, congenital immunodeficiency disorders, or organ transplantation history;
* The baseline pregnancy test was positive for pregnant, lactating or fertile women, and the patients of childbearing age who were unwilling to take effective contraceptive measures during the whole period of the test were unwilling to take effective contraceptive measures;
* According to the judgement of researchers, there are concomitant diseases that seriously endanger patients'safety or affect patients' completion of research;
* There was a clear history of neurological or psychiatric disorders, including epilepsy or dementia;
* Researchers believe that patients are not suitable for any other situation in this study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 5 month
  Progression free survival

SECONDARY OUTCOMES:
OS | through study completion, an average of 18 month
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yongqian Shu, professor, Study Chair — JANGSU PROVINCE HOSPITAL
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu Y, Miao L, Chen X, Zhu X, Li Y, He J, Chen P, Dai S, Liu Z, Ma K, Wang N, Zhao Y, Chen N, Song W, Bai R, Cui J, Shu Y. Maintenance therapy with anlotinib after induction therapy with platinum-based chemotherapy for advanced non-small-cell lung cancer: A pooled analysis of 2 single-arm trials. Medicine (Baltimore). 2024 Jul 5;103(27):e38459. doi: 10.1097/MD.0000000000038459. PMID 38968520